CLINICAL TRIAL: NCT04852822
Title: Multicenter Evaluation of SARS-CoV-2 Vaccines in Patients With CLL/SLL
Brief Title: Immune Response to SARS-CoV-2 (COVID-19) Vaccines in Patients With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Terminated | Type: Observational
Why Stopped: The study ended earlier than anticipated due to slow accrual.
Sponsor: University of Washington (Other)
Collaborators: CLL Global Research Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: RG1121418; NCI-2021-02178 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10646 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2021-04-19; First posted 2021-04-21 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, medical record review): For patients who have not been vaccinated at the time of enrollment, they will undergo collection of blood samples prior to the first vaccine dose, just before the second vaccine dose, and then at 1, 6, and 12 months after the second vaccine dose. Patients' medical records are also reviewed.
  For patients enrolled after vaccination, they will undergo collection of blood samples at 1-4, 6, and 12 months after completing the vaccination series. Patients who receive booster dose also undergo collection of blood samples at 1, 6, and 12 months post final booster dose.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
Other: Electronic Health Record Review — Medical records are reviewed

SUMMARY:
This study evaluates the immune response to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccines in patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL). CLL and SLL are types of blood cancer that begin in cells of the immune system. CLL/SLL and the medications used to treat these conditions may change the way vaccines work in a patient's body. The purpose of this study is to find out if patients with CLL/SLL make antibodies, or have an immune response, to the SARS-CoV-2 vaccines. Information gained from this study may help researchers better understand how effective the vaccines work in preventing COVID-19 (coronavirus disease 2019) in patients with CLL and SLL.

DETAILED DESCRIPTION:
OUTLINE:

For patients who have not been vaccinated at the time of enrollment, they will undergo collection of blood samples prior to the first vaccine dose, just before the second vaccine dose, and then at 1, 6, and 12 months after the second vaccine dose. Patients' medical records are also reviewed.

For patients enrolled after vaccination, they will undergo collection of blood samples at 1-4, 6, and 12 months after completing the vaccination series. Patients who receive booster dose also undergo collection of blood samples at 1, 6, and 12 months post final booster dose.

After completion of study, patients are followed up every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* A diagnosis of chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL)
* Willing and able to participate in all required evaluations and procedures in this study

Exclusion Criteria:

* Any evidence of prior SARS-CoV-2/COVID19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) who receive a SARS-CoV-2 vaccine
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Response rate to the SARS-CoV-2 vaccine among patients with chronic lymphocytic leukemia/small lymphocytic lymphoma | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chaitra S. Ujjani, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (11):
- United States (11):
  - City of Hope, Duarte, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ujjani C, Gooley TA, Spurgeon SE, Stephens DM, Lai C, Broome CM, O'Brien S, Zhu H, Laing KJ, Winter AM, Pongas G, Greninger AL, Koelle DM, Siddiqi T, Davids MS, Rogers KA, Danilov AV, Sperling A, Tu B, Sorensen T, Launchbury K, Burrow CJ, Quezada G, Hill JA, Shadman M, Thompson PA. Diminished humoral and cellular responses to SARS-CoV-2 vaccines in patients with chronic lymphocytic leukemia. Blood Adv. 2023 Sep 12;7(17):4728-4737. doi: 10.1182/bloodadvances.2022009164. PMID 36516082

DOCUMENTS (1):
  • Informed Consent Form (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT04852822/ICF_000.pdf